CLINICAL TRIAL: NCT04151940
Title: An Interventional Study of PET/CT Changes During Chemoimmunotherapy and Radiation Therapy for Patients With Metastatic NSCLC (PET Bright)
Brief Title: PET/CT Changes During Chemoimmunotherapy and Radiation Therapy in Patients With Stage IV Non-small Cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RG1005458; NCI-2019-07068 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10203 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA258997 (NIH)
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
Keywords: Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Magnetic Resonance Spectroscopy; X-Rays; Drug Therapy; Immunotherapy; Adjuvants, Immunologic; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Research (PET/CT scan) (Experimental): Patients undergo PET/CT scan within 4 weeks before starting standard of care chemoimmunotherapy and a second PET/CT scan within 5 days of the second chemoimmunotherapy cycle. Patients receiving standard of care radiation treatment undergo additional PET/CT scans within 4 weeks prior to radiation treatment and 1 month post-radiation treatment. Additionally, patients undergo blood sample collection on study. Patients may also undergo MRI as clinically indicated throughout the study.
  Interventions: Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Drug: Chemotherapy; Biological: Immunotherapy; Radiation: Radiation Therapy; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging; PET; PET scan; positron emission tomography scan; Positron-Emission Tomography; PT
Procedure: Computed Tomography — Undergo PET/CT scan
  Other Names: CAT; CAT Scan; computerized axial tomography; computerized tomography; CT; CT SCAN
Drug: Chemotherapy — Receive standard of care chemotherapy
  Other Names: Chemo; Chemotherapy (NOS)
Biological: Immunotherapy — Receive standard of care immunotherapy
  Other Names: Immunological; Immunological Therapy; Immunologically Directed Therapy
Radiation: Radiation Therapy — Undergo standard of care radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; irradiated; Irradiation; Radiation; Radiotherapeutics; radiotherapy; RT
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI; MRI Scan

SUMMARY:
This study investigates the changes in positron emission tomography (PET)/computed tomography (CT) imaging scans during chemoimmunotherapy and radiation therapy treatment in patients with stage IV non-small cell lung cancer. Analyzing changes in PET/CT imaging scans may help doctors assess and predict patterns of cancer response to chemoimmunotherapy and radiation therapy.

DETAILED DESCRIPTION:
Patients undergo PET/CT scan within 4 weeks before starting standard of care chemoimmunotherapy and a second PET/CT scan within 5 days of the second chemoimmunotherapy cycle. Patients receiving standard of care radiation treatment undergo additional PET/CT scans within 4 weeks prior to radiation treatment and 1 month post-radiation treatment. Additionally, patients undergo blood sample collection on study. Patients may also undergo magnetic resonance imaging (MRI) as clinically indicated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed or cytologically-confirmed metastatic NSCLC in patients who have not received chemotherapy or immunotherapy for their advanced disease (stage IV or recurrent, using the American Joint Committee on Cancer [AJCC]/Union for International Cancer Control [UICC] 8th edition for staging)
* Evidence of stage IV disease on imaging by CT, PET/CT, or magnetic resonance imaging (MRI)
* Plan to treat with a platinum doublet with a PD1 or PDL1 inhibitor
* Adjuvant chemotherapy or concurrent chemoradiation for early stage disease does not count as prior therapy unless subject progressed within 6 months of completion of regimen.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1, at treating physician's discretion
* Subjects must be ≥ 18 years of age
* Patients with known activating mutations in EGFR, BRAF or known translocation in ALK or ROS-1 are eligible provided they have progressed on or were intolerant to Food and Drug Administration (FDA) approved targeted therapy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Creatinine =< 2 mg/dL or creatinine clearance > 50 mL/min
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5x institutional upper limit of normal
* Total bilirubin =< 1.5 mg/dL
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (>= 1500 per mm^3)
* Platelet count >= 100 x 10^9/L (>=100,000 per mm^3)
* Capability to understand and comply with the protocol requirements and signed informed consent documents

Exclusion Criteria:

* Any known additional malignancy (with exception of non-melanoma skin cancer, in-situ breast cancer, low risk prostate cancer, or a malignancy diagnosed >= 3 years prior to the current NSCLC diagnosis and with no evidence of requiring active treatment)
* Had prior treatment with an anti-PD-1, or PD-L1 or PD-L2 agent or an antibody targeting other immuno-regulatory receptors or mechanisms
* Has any serious or uncontrolled active infection that could create false positives on a PET/CT scan, in the opinion of the treating investigator
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has an active autoimmune disease currently requiring systemic treatment (e.g. disease modifying agents, corticosteroids or immunosuppressive drugs)

  **Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known, active, and symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis

  * Patients with stable or previously treated brain metastases are eligible as long as they are not receiving more than 10 mg of prednisone, or equivalent, per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Actuarial disease progression rate | At 1 year
  Will be compared between high-risk and low-risk subgroups of patients based on positron emission tomography/computed tomography imaging biomarker changes using a two-sample proportionality test.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Deng, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No